CLINICAL TRIAL: NCT03685162
Title: Observational, Prospective Study to Evaluate Levomethadone Safety Profile and Effectiveness in Subjects Under Opioid Maintenance Treatment
Brief Title: Observational Study to Evaluate Levomethadone Safety and Effectiveness in Subjects Under Opioid Maintenance Treatment
Acronym: LEVOPROACT
Status: Completed | Type: Observational
Sponsor: L.Molteni & C. dei F.lli Alitti-Soc. di Esercizio S.p.A. (Industry)
Responsible Party: Sponsor
Other Study IDs: MOLT-2015-01
Record Dates: First submitted 2018-04-17; First posted 2018-09-26 (Actual); Last update posted 2023-10-24 (Actual); Status verified 2023-10

CONDITIONS: Opioid Addiction
Keywords: addiction; opioid addiction; levomethadone; methadone; opioid maintenance treatment
MeSH Terms: conditions — Opioid-Related Disorders; Behavior, Addictive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

SUMMARY:
Multicentre, prospective, observational, non-interventional, open- ended trial, collecting data from male and female patients aged ≥ 18 years, with a diagnosis of opioid addiction according to ICD-10 (F11.2), treated with therapeutic doses of levomethadone according to the routine medical practice.

DETAILED DESCRIPTION:
Multicentre, prospective, observational, non-interventional, open- ended trial, collecting data from male and female patients aged ≥ 18 years, with a diagnosis of opioid addiction according to ICD-10 (F11.2), treated with therapeutic doses of levomethadone according to the routine medical practice.

The study is divided in two different consecutive parts:

* Part 1 [from Informed Consent form (ICF) to last data collected at V4]: patients enrolled are receiving levomethadone maintenance treatment according to clinical practice.
* Part 2 (after V4 up to FU): patients are in opioid maintenance treatment with any drug (including levomethadone) according to clinical practice.

The maximum duration on-study for a patient will be 405 days [from ICF signature (-30 days from V1) to FU (=360 + 15)]. This study is an open-ended trial. This means that for the enrolment and for the study, no maximum duration has been established.

The study, which is a voluntary Post Authorization Safety Study (PASS), will be carried out on approximately 10 centers in Italy.

The objectives are to provide further data on the safety profile after long term use and effectiveness of levomethadone, administered according Summary of Product Characteristics (SmPC) and in a real word clinical setting, in opioid-addicted patients undergoing maintenance treatment.

Safety will be assessed throughout all the study and safety data will be described and analysed based on Adverse Drug Reactions and corrected QT (QTc) prolongation at 12-lead electrocardiogram (ECG), where available.

The effectiveness outcomes are the evaluation of levomethadone maintenance treatment according to investigator's judgment at V4(180 days), based on different questionnaires and assessment.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients, aged ≥ 18 years;
* Patients with a diagnosis of opioid addiction according to ICD-10 (ICD 10 F11.2);
* Opioid-addicted patients initiating or currently undergoing a maintenance treatment with levomethadone as part of their routine clinical care and according to the approved SmPC;
* Patients or legal guardian when applicable must provide their written informed consent to participate in the study.

Exclusion Criteria:

* Inability to understand study procedures;
* Any contraindication stated in the SmPC for the administration of levomethadone according to investigator's judgment;
* Patients currently participating in any other clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female patients aged ≥ 18 years, with a diagnosis of opioid addiction according to ICD-10 (F11.2), treated with therapeutic doses of levomethadone according to the routine medical practice.
Sampling Method: Probability Sample
Enrollment: 103 (Actual)
Dates: Start 2018-02-27 (Actual); Primary Completion 2023-02-16 (Actual); Study Completion 2023-02-16 (Actual)

PRIMARY OUTCOMES:
Safety (based on Adverse Drug Reactions) | Safety will be described throughout all the study (maximum duration approximately 1 year).
  Safety will be assessed throughout all the study and safety data will be described and analysed based on Adverse Drug Reactions.
Effectiveness (Addiction Severity) | The effectiveness outcomes will be evaluated at V4 (180 days).
  Assessed by Addiction Severity Index (ASI); ASI is a semi-structured interview that consent to assess addiction severity (scale 0-9; 0: no problems, 9: severe problems) of the patient in 7 problem areas.
Effectiveness (Substance use) | The effectiveness outcomes will be evaluated at V4 (180 days).
  The patient will register on a diary the use (days) of heroin, buprenorphine, cocaine.
Effectiveness (Presence of Catabolites) | The effectiveness outcomes will be evaluated at V4 (180 days).
  Assessment (negative/positive) of heroin, methadone, buprenorphine, cocaine in urine.
Effectiveness (Retention Rate) | The effectiveness outcomes will be evaluated at V4 (180 days).
  Retention rate (days) in treatment with levomethadone.
Effectiveness (Craving) | The effectiveness outcomes will be evaluated at V4 (180 days).
  Craving will be assessed using by Visual Analogue Scale (VAS) (0-100mm; 0: no craving, 100: maximum craving)
Effectiveness (Evaluation of Quality of life) | The effectiveness outcomes will be evaluated at V4 (180 days).
  The evaluation of quality of life will be carried out with the Quality of Life Short-Form Health Survey questionnaire (SF-12). This questionnaire takes into account two domains: Physical Component Summary (PCS-12) and Mental Component Summary (MCS-12) where the lower the score the more disability and the higher the score the less disability.

CONTACTS AND LOCATIONS:
Locations (1):
- UOC Dipendenze, ASST Papa Giovanni XXIII, Bergamo, Italy